CLINICAL TRIAL: NCT04148417
Title: Clinical Study of the Solo+ Tympanostomy Tube Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AventaMed DAC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP002
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Ear Infection; Otitis Media
MeSH Terms: conditions — Otitis; Otitis Media

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Solo+ Tympanostomy Tube Device (Experimental): The Solo+ Tympanostomy Tube Device is a disposable surgical tool designed to deliver a tympanostomy tube (grommet) into the tympanic membrane of patients undergoing a tympanostomy tube placement procedure
  Interventions: Device: Solo+ Tympanostomy Tube Device

INTERVENTIONS:
Device: Solo+ Tympanostomy Tube Device — The Solo+ Tympanostomy Tube Device is intended to deliver a tympanostomy tube through the tympanic membrane of a patient during a tympanostomy procedure

SUMMARY:
The objective of this study is to evaluate the safety and performance of the Solo+ Tympanostomy Tube Device for the placement of tympanostomy tubes (grommets) in paediatric patients undergoing a tympanostomy procedure

DETAILED DESCRIPTION:
The study will be a multi-site, prospective, treatment-only study of the Solo+ Tympanostomy Tube Device. Patients will already have a scheduled tympanostomy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Listed for bilateral tympanostomy tube insertion

Exclusion Criteria:

* Anatomy that precludes sufficient visualisation of both the left and right eardrum
* Narrow ear canals
* Anatomy that precludes safe access to both the left and right eardrum
* Membrane >25% sclerosis
* Congenital or craniofacial abnormalities
* No available baseline audiometry and tympanometry

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Successful delivery of the tympanostomy tube by the Solo+ Tympanostomy Tube Device | Intra-operative
  The number of ears in which the Solo Tympanostomy Tube Device tube is placed
Rate of Adverse Events | 24 months
  The number and type of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Matija Daniel, Study Chair — Queen's Medical Center
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No